CLINICAL TRIAL: NCT03111615
Title: Hormone Therapy Initiation Immediately After Histological Diagnosis of Breast Cancer, Can it Make Any Difference?
Brief Title: HOrmone Therapy Immediately After Histological Diagnosis of Breast Cancer
Acronym: HOTBreast
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Hospitalar Lisboa Ocidental (Other Government)
Responsible Party: Principal Investigator, Zacharoula Sidiropoulou, Principal investigator, Centro Hospitalar Lisboa Ocidental
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CentroHLOBreastUnit
Record Dates: First submitted 2017-02-23; First posted 2017-04-13 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Hormone Dependent Neoplasms; Breast Cancer Female
Keywords: Aromatase inhibitors; Luminal Breast Cancer neoadjuvant hormone therapy
MeSH Terms: conditions — Neoplasms, Hormone-Dependent | interventions — Aromatase Inhibitors

STUDY DESIGN:
Intervention Model Description: Aromatase inibitor therapy to start immediately after biopsy results are available Letrozole 2.5mg or Anastrazol 1 mg
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aromatase Inhibitor group (Experimental): Female patients of 50 and above y.o. shall initiate hormone therapy (Letrozol 2.5 mg or Anastrazol 1 mg) immediately after the diagnosis until surgery.
  Interventions: Drug: Aromatase Inhibitors
- Control group (No Intervention): Female patients of 50 and above y.o. that follow standard protocol (no pre-surgery (Letrozol 2.5 mg or Anastrazol 1 mg))
- Aromatase Inhibitor Active surveillance (Other): Female patients of 50 and above y.o. that refuse surgery and therefor follow standard protocol (only Letrozol 2.5mg or Anastrazol 1 mg) until disease progression, death or will of surgery In this subgroup we are going to include, under HT, female patients with CDis,that refuse the standard treatment with surgery plus eventual rt and/or ht
  Interventions: Drug: Aromatase Inhibitors
- Aromatase Inhibitor Active surveillance + aas (Other): emale patients of 50 and above y.o. that refuse surgery and therefor follow standard protocol (only Letrozol 2.5mg or Anastrazol 1 mg plus acetilsalicilic acid) until disease progression, death or will of surgery In this subgroup we are going to include, under HT, female patients with CDis,that refuse the standard treatment with surgery plus eventual rt and/or ht
  Interventions: Drug: Aromatase Inhibitors

INTERVENTIONS:
Drug: Aromatase Inhibitors — Aromatase Inhibitor to start immediately after diagnosis of a Luminal Invasive Breast Carcinoma Patients will be given Letrozol 2.5 mg or Anastrazol1 mg, every 24H and all of them will be given Calcium + Vit D supplement.
  Venlafaxin 75 mg is to be administrated cases indicated
  Other Names: Aromatase Inhibitor
  Arms: Aromatase Inhibitor Active surveillance; Aromatase Inhibitor Active surveillance + aas; Aromatase Inhibitor group

SUMMARY:
Breast Cancer is a public health issue worldwide. The time from diagnosis to treatment initiation varies from country to country and regionally within a country. Early diagnosis and prompt treatment initiation are key factors in patient survival rates.

Currently there is a rising trend, with a high percentage of patients with "Luminal" like breast cancer only undergoing adjuvant endocrine therapy.

Authors argue that tumor biology alterations after introducing very early endocrine therapy might have a prognostic and therapeutic impact and should be studied.

DETAILED DESCRIPTION:
Selected patients of female gender, above 50 y.o, and after a biopsy of Luminal-like Breast Cancer will go under aromatase inhibitor, from the diagnosis day till the surgical therapy to be decided (if so).In this study are going to be included patients that refuse surgical treatment, remaining this way in an "active surveillance". This last group is going to be randomised in order to recieve hormontherapy plus placebo vs hormontherapy plus acetolisalicilic acid.

In this way, authors want to investigate if:

1. st This approach influences the tumor biology
2. nd This approach influences tumor pathologic response and progression free survival.
3. rd It is a valid approach and in which grade, for patients that refuse surgical treatment

ELIGIBILITY:
Inclusion Criteria: Menopausal woman of equal or above 50 y.o. with breast biopsy of Luminal like breast carcinoma

Exclusion Criteria:

* informed consent
* <50 y.o.
* Pre-menopausal state

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female sex
Enrollment: 90 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Tumor Biology | 6 weeks
  Effects of neoadjuvant aromatase inibitors on tumor biology in terms of RE,PR,Ki 67 measuring the after IA presurgical values

SECONDARY OUTCOMES:
Tumor Pathology response | 6 weeks
  Effects of neoadjuvant aromatase inibitors on tumor pathologic response , in terms of breast imaging re-avaliation before surgical intervention. For patients that refuse surgery or extend hormone therapy for other reasons
Disease free survival | 1 5 and 10 years
  Effects of neoadjuvant aromatase inibitors on disease free survival the first, fifth and tenth years of follow-up
Hormone treatment | 1 5 and 10 years
  Disease stability or progression under Hormone treatment in patients under active surveillance. Clinical and immaging follow up

OTHER OUTCOMES:
Surgical outome | 3 days 1 month and 3 months
  Eventual influence of the aromatase inibitor in the surgical procedure (time, bleeding, scaring, infections, seroma formation, sentinel node detection and axillary response) is to be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Vasco Fonseca, MD, Principal Investigator — CHLO Medical Oncology dpt; Zacharoula Sidiropoulou, Principal Investigator — CHLO Surgery dpt
Locations (1):
- Hospital São Francisco Xavier, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No